CLINICAL TRIAL: NCT03652168
Title: Stress Free UC Merced: The Effect of 8 Weeks of Mindfulness App Headspace on Stress in a Sample of University Employees
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, Merced (Other)
Collaborators: The University of California's Healthy Campus Network (Other); Headspace Meditation Limited (Industry)
Responsible Party: Principal Investigator, Matthew Zawadzki, Assistant Professor, University of California, Merced
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCM2018-9
Record Dates: First submitted 2018-08-17; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Stress; Psychological Distress
Keywords: stress; health; mindfulness; employees
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The party or parties involved in the clinical trial who are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): Headspace application: Participants in the intervention group will use a digitally-based mindfulness intervention Headspace app (Basics + Stress packs) will be used for 10 minutes a day over the course of 8 weeks.
  Interventions: Behavioral: Meditation
- No intervention, control group (No Intervention): Control group participants will continue their normal activities and not add any form of meditation during the study period.

INTERVENTIONS:
Behavioral: Meditation — 10 minute a day, 8 week digital meditation
  Arms: Meditation Group

SUMMARY:
The aim of this study is to investigate the effects of the app-based mindfulness intervention (i.e., the commercially available application Headspace) on overall physical and psychological health. Secondly, this study examines potential mindfulness mechanisms that may be driving these effects (i.e., decentering, attention regulation, acceptance, self-compassion, reactivity, exposure).

This study will randomize UC Merced employees to 8-weeks of either a digital mindfulness intervention (Headspace) or a waitlist control condition. Participants assigned to the intervention group will be asked to download and use the Headspace mobile application for 10 minutes per day for 8 weeks. They will be asked to fill out questionnaires at baseline, week 4, week 8 (post intervention), 4-month, and 12-month follow up period (20-30 minutes each time). In addition, participants will be asked to complete surveys on their phone as a part of everyday life assessments (4 days per week during baseline, 2 weeks, 5 weeks, 8 weeks, up to 5-10 minutes a day). Participants will also wear a fitness watch, Fitbit, to assess their activity, sleep, and heart rate data. For the everyday life assessment part, participants will be asked to participate in one of our 60 minutes orientation sessions where you will receive training on using the mobile app and receive a fitness watch that will be collected upon the completion of the study.

DETAILED DESCRIPTION:
Stress at work has shown to be an important health risk for employees. It is associated with poor mental and physical health including anxiety, depression, sleep disturbances, gastrointestinal problems, type 2 diabetes, and cardiovascular disease. Work stress also has major implications for employers as evidence suggests that high levels of work stress predict employee burnout, turnover intent, absenteeism, and poor job performance.

Mindfulness and its positive effects on a variety of outcomes, including stress reduction, have been documented in many studies. The most common definition of mindfulness is as the state of being attentive to and aware of the present moment with an attitude of openness and acceptance. Several mechanisms by which mindfulness exerts its positive effects have been proposed in the literature including cultivating the attitude of non-judgement and acceptance, ability to observe one's experiences objectively without reacting to them, and ability to be more patient and kind toward oneself. Recent evidence suggests that teaching mindfulness in the workplace not only reduces stress but also improve psychological well-being.

With advances in technology, technology-based delivery of many interventions has become popular. App-based treatments for improving psychological health are becoming increasingly important due to high accessibility and cost-effectiveness of smartphone technology. Despite a great number of app-based interventions, there has been little research evaluating their efficacy. Support for the use of smartphone app-based mindfulness interventions comes from a few small studies that found these interventions to produce benefits comparable to traditional delivery methods. While app-based interventions offer a convenient alternative to traditional delivery methods as well as promising initial empirical evidence, more research is needed in order to further evaluate and promote these interventions.

The proposed study has several goals. The first goal is to investigate the effects of the app-based mindfulness intervention on overall physical and psychological health (e.g., perceived stress, mindfulness, sleep quality, self-reported health, anxiety symptoms). The second goal is to examine the effect of the intervention on a variety of work-related outcomes (e.g., work stress, job satisfaction, work-related burnout). Further, the study will examine potential mindfulness mechanisms that may drive these effects (e.g., acceptance, reactivity, decentering).

ELIGIBILITY:
Inclusion Criteria:

* Have access to a smartphone or computer with internet every day
* Are fluent in English
* Are a UC Merced employee
* Consent: demonstrate understanding of the study and willingness to participate as evidenced by voluntary informed consent and has received a signed and dated copy of the informed consent
* Are at least 18 years of age

Exclusion Criteria:

* Individuals may not join if they are experienced meditators or have participated in a sitting meditation practice more than twice a week (for 10 minutes or greater) over the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
10-Item Measure of Stress Perceptions | Change from Baseline Stress Perceptions at 12 months
  Self-reported stress perceptions over the over the past month. Each item is scored using a 0 (never) and 4 (very often) scale. Items are averaged together such that scores can range from 0 to 40; higher scores indicate higher perceived stress. Total score ranging from 0-13 would be considered low stress. Score ranging from 14-26 would be considered moderate stress. Score ranging from 27-40 would be considered high perceived stress.

SECONDARY OUTCOMES:
9-Item Measure of Symptoms of Depression and Distress | Change from Baseline Depression at 12 months
  Self-reported symptoms of depression and distress over the last two weeks. Answers range from 0 (not at all) to 4 (nearly every day). Scores are added across columns to get a total score. Scores can range from 0 to 36, the lowest score of 1- 4 indicate minimal depression; higher scores 20-27 indicating severe depression.
7-Item Measure of Symptoms of Anxiety | Change from Baseline Anxiety at 12 months
  Self-reported symptoms of anxiety over the last two weeks. Answers range from 0 (not at all) to 4 (nearly every day). Scores are added across columns to get a total score. Scores can range from 0 to 28 and scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
15-Item Measure of Mindfulness - a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present | Change from Baseline Mindfulness at 12 months
  Self-reported mindfulness ratings participants report on average each day. Answers are given on a 1 (almost always) to 6 (almost never) scale. Total score is calculated by computing a mean of the 15 items. Scores can range from 15 to 90 with higher scores reflect higher levels of dispositional mindfulness.
19-Item Measure of Sleep Quality | Change from Baseline Sleep Quality at 8 weeks
  Self-reported measure of sleep quality over the last month. The self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a total score of "0" indicates no difficulty and "21" indicating severe difficulties in all areas.
1-Item Measure of Leisure Physical Activity | Change from Baseline Physical Activity at 8 weeks
  Self-reported measure of physical activity performed on average during leisure activity over the past month. Item is scored on a 0 (no physical activity) to 4 (vigorous activity at least 3 times a week) scale
Resting Heart Rate | Change from Baseline Resting Heart Rate at 8 weeks
  The Fitbit watch worn during the intervention will assess resting heart rate levels each day.
12-Item Subjective Mental and Physical Well-Being Ratings | Change from Baseline Self-reported health at 8 weeks
  Self-reported measure of views about mental and physical well-being on average. The items are scored on a 0 to 100 and averaged, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
3-Item Job Satisfaction Measure | Change from Job Satisfaction at 12 months
  Self-reported assessment of average levels of job satisfaction. Items are scored on a 1 (Disagree very much) to 6 (Agree very much) with an average total score across items ranging from 3 to 18.
5-Item Work-Family Balance Measure of emotional, behavioral and time demands of both paid work and family (if relevant) or personal duties. | Change from Baseline Work-family Balance at 12 months
  Self-reported measure of work-family balance on average. Items are scores on a 1 (strongly disagree) to 7 (strongly agree) scale. Items are averaged together with the total score ranging from 5 to 35.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Zawadzki, PhD, Principal Investigator — UC Merced
Locations (1):
- University of California, Merced, Merced, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bishop, S. R., Lau, M., Shapiro, S., Carlson, L., Anderson, N. D., Carmody, J., ... & Devins, G. (2004). Mindfulness: A proposed operational definition. Clinical psychology: Science and practice, 11(3), 230-241.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Ganster, D. C., & Rosen, C. C. (2013). Work stress and employee health: A multidisciplinary review. Journal of Management, 39(5), 1085-1122.
- [Background] Goedhard, R. G., & Goedhard, W. J. (2005, June). Work ability and perceived work stress. In International Congress Series(Vol. 1280, pp. 79-83). Elsevier.
- [Background] Jamieson SD, Tuckey MR. Mindfulness interventions in the workplace: A critique of the current state of the literature. J Occup Health Psychol. 2017 Apr;22(2):180-193. doi: 10.1037/ocp0000048. Epub 2016 Sep 19. PMID 27643606
- [Background] Fairburn CG, Patel V. The impact of digital technology on psychological treatments and their dissemination. Behav Res Ther. 2017 Jan;88:19-25. doi: 10.1016/j.brat.2016.08.012. PMID 28110672
- [Background] Howells, A., Ivtzan, I., & Eiroa-Orosa, F. J. (2016). Putting the 'app'in happiness: a randomised controlled trial of a smartphone-based mindfulness intervention to enhance wellbeing. Journal of Happiness Studies, 17(1), 163-185.